CLINICAL TRIAL: NCT01696773
Title: Enhancing Bioavailability and Nutritional Quality of Processed Tomato Products
Brief Title: Carotenoid and Flavonoid Absorption From Red and Tangerine-Type Tomatoes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jessica Cooperstone, Assistant Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2012H0189
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Carotenoid and Flavonoid Absorption
Keywords: tomato; tangerine tomato; carotenoids; lycopene; flavonoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tangerine tomato juice (Experimental): Tangerine tomato juice will be fed
  Interventions: Other: Tangerine tomato juice
- Red tomato juice (Experimental): Red tomato juice will be fed
  Interventions: Other: Red tomato juice

INTERVENTIONS:
Other: Tangerine tomato juice — Post-prandial feeding study
  Arms: Tangerine tomato juice
Other: Red tomato juice — Post-prandial feeding study
  Arms: Red tomato juice

SUMMARY:
Eating a diet rich in tomatoes has been associated with decreased risk for a variety of diseases. Tomatoes contain red-colored lycopene (one type of pigment in the class of pigments called carotenoids), which has been associated with the decreased risk of disease in those consuming tomato products; however, tomatoes also contain flavonoids, which may also have health promoting effects. The Tangerine tomato, a unique tomato variety, contains lycopene in a different form that in red tomatoes and this contributes to their characteristic orange color. This "orange lycopene" is more similar to the most common form of lycopene found in the blood and tissue of people who eat a tomato-rich diet, and may be more easily absorbed by the body.

The objectives of this study are to determine if carotenoids and flavonoids from Tangerine tomatoes are more easily absorbed by the body than red tomatoes, and to examine if eating Tangerine versus red tomatoes impacts markers of inflammation (response to harmful substances by the body).

DETAILED DESCRIPTION:
The primary goal of this research is to determine if a processed Tangerine tomato product has enhanced bioavailability of carotenoids and flavonoids compared to a commercially available processed red tomato product in humans. This primary objective will be accomplished by quantifying carotenoids from post-prandial triglyceride-rich lipoprotein (TRL) fractions of plasma and flavonoids from whole plasma and urine, after subjects consume a meal containing Tangerine or red tomato juice. A secondary goal is to examine if short-term delivery of bioactives from Tangerine and red tomatoes impact markers of inflammation in humans. This secondary objective will be accomplished by analyzing plasma for both interleukin-6 (IL-6), a marker for inflammation, and RNA to assess alterations in transcription of genes that regulate inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Total cholesterol ≤200 mg/dL
* Triglycerides ≤ 200mg/dL
* BMI 18.5 to 30.0kg/m2
* Not anemic (hemoglobin at or above 10g/dL and hematocrit at or above 30%)
* Age 18-70 years

Exclusion Criteria:

* Lactating, pregnant, or plan to be pregnant during study
* Tobacco (cigarettes and chewing tobacco)
* Metabolic disease, such as diabetes mellitus or thyroid dysfunction
* Malabsorption disorders (e.g. ileus, Crohn's, ulcerative colitis, pancreatic insufficiency)
* History of cancer, esophageal, gastric, or intestinal ulcers
* History of liver or kidney insufficiency or failure
* Auto-immune disorders
* Chronic inflammation (e.g. rheumatoid arthritis)
* Allergies to tomatoes or tomato products
* Obesity (BMI > 30kg/m2) or underweight (BMI <18.5kg/m2)
* Hypercholesterolemia (Total cholesterol > 200 mg/dL)
* Triglycerides > 200mg/dL
* Subjects taking non-steroidal anti-inflammatory medications (e.g. Aspirin, Advil, Tylenol, Aleve) for 72 hours prior to each day-long visit.
* Anemia (hemoglobin below 10g/dL or hematocrit below 30%)
* Blood donation within the last 8 weeks

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2027-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Schwartz, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Clinical Research Center, Columbus, Ohio, United States

REFERENCES:
- [Derived] Cooperstone JL, Ralston RA, Riedl KM, Haufe TC, Schweiggert RM, King SA, Timmers CD, Francis DM, Lesinski GB, Clinton SK, Schwartz SJ. Enhanced bioavailability of lycopene when consumed as cis-isomers from tangerine compared to red tomato juice, a randomized, cross-over clinical trial. Mol Nutr Food Res. 2015 Apr;59(4):658-69. doi: 10.1002/mnfr.201400658. Epub 2015 Mar 10. PMID 25620547

RESULTS

PARTICIPANT FLOW:
Groups:
- Tangerine Tomato Juice First, Then Red Tomato Juice: Tangerine tomato juice will be fed, followed by a 14 day washout, and then red tomato juice will be fed
- Red Tomato Juice First, Then Tangerine Tomato Juice: Red tomato juice will be fed, followed by a 14 day washout, then tangerine tomato juice will be fed.
Period: Days 1-13, Washout
Arm/Group | Tangerine Tomato Juice First, Then Red Tomato Juice | Red Tomato Juice First, Then Tangerine Tomato Juice
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Day 14, First Intervention
Arm/Group | Tangerine Tomato Juice First, Then Red Tomato Juice | Red Tomato Juice First, Then Tangerine Tomato Juice
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Days 15-27, Washout
Arm/Group | Tangerine Tomato Juice First, Then Red Tomato Juice | Red Tomato Juice First, Then Tangerine Tomato Juice
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Day 28, Second Intervention
Arm/Group | Tangerine Tomato Juice First, Then Red Tomato Juice | Red Tomato Juice First, Then Tangerine Tomato Juice
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tangerine Tomato Juice First, Then Red Tomato Juice: Tangerine tomato juice is consumed on day 14 then red tomato juice on day 28
- Red Tomato Juice First, Then Tangerine Tomato Juice: Red tomato juice is consumed on day 14, then tangerine tomato juice on day 28
- Total: Total of all reporting groups
Arm/Group | Tangerine Tomato Juice First, Then Red Tomato Juice | Red Tomato Juice First, Then Tangerine Tomato Juice | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.8 (2.8) | 29.0 (13.4) | 25.9 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
BMI [Mean (Standard Deviation); unit: kg/m^2] | 23.1 (1.4) | 25.5 (1.6) | 23.3 (1.4)
Plasma cholesterol (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 170.6 (8.9) | 176.2 (12.5) | 173.8 (10.6)
Plasma triglycerides (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 65.8 (49.3) | 85.8 (42.3) | 75.8 (45.0)
Hematocrit [Mean (Standard Deviation); unit: Volume % of red blood cells in blood] | 41.8 (2.8) | 42.0 (3.8) | 41.9 (3.2)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 13.9 (0.8) | 14.1 (1.1) | 14.0 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Carotenoid Absorption
Description: The primary goal of this research is to determine if a processed tangerine tomato product has enhanced bioavailability of carotenoids and flavonoids compared to a commercially available processed red tomato product in humans. An area under the curve for concentration of carotenoids (from triglyceride rich lipoprotein (TRL) fraction of plasma) by using carotenoid concentrations from hours 0, 2, 3, 4, 5, 6, 8, 10 and 12 over time to quantify absorption, after subjects consume a meal containing tangerine or red tomato juice.
Time Frame: 11 post-prandial blood samples will be taken over 12 hours
Measure: Mean (Standard Error); unit: nmol*h/L
Arm/Group | Tangerine Tomato Juice | Red Tomato Juice
Number analyzed (Participants) | 11 | 11
nmol*h/L | 690.9 (117.8) | 81.6 (32.1)

ADVERSE EVENTS:
Arm/Group | Tangerine Tomato Juice | Red Tomato Juice
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 1/12 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tangerine Tomato Juice (N=12) | Red Tomato Juice (N=11)
Menstrual distress (Reproductive system and breast disorders) | 1 (1) | 0 (0) — 1 subject chose to dropout of the study 4 days after the first day long visit (at day 18). Adverse event categorized as sexual/reproductive function - other, menstrual distress - mild to moderate, not attributable or associated with the study agent.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No